CLINICAL TRIAL: NCT05477251
Title: Comparative Study on the Efficacy and Safety of Microwave Ablation and Lobectomy in the Treatment of Ground Glass Nodules Located in the Pulmonary Hilar Region
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Chi Jiachang, Deputy Chief Physician, RenJi Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2021-263-B
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Pulmonary Nodule, Multiple; Pulmonary Nodule, Solitary
MeSH Terms: conditions — Multiple Pulmonary Nodules; Solitary Pulmonary Nodule | interventions — Anterior Temporal Lobectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- microwave ablation (Experimental)
  Interventions: Procedure: microwave ablation
- lobectomy (Active Comparator)
  Interventions: Procedure: lobectomy

INTERVENTIONS:
Procedure: microwave ablation — MWA procedures were performed under local anesthesia and CT guidance (GE Discovery CT750 HD) was used for the guidance. Using the coaxial system, MWA was performed by the combining of a 17G sharp-tip guide trocar needle and a 15-cm cooled-shaft electrode (18-gauge) with a 1.5-cm expandable blunt-tip (MTC-3CA-II3, Vison Medical Inc.). Firstly, the sharp-tip guide trocar needle was used to puncture through the pleura and then the blunt-tip MWA electrode was advanced into the GGO lesion through the guide needle lumen. Once the target was reached, ablation was performed at a power of 40 watts. Once the lesion was covered by the ablation zone, the ablation completed.
  Arms: microwave ablation
Procedure: lobectomy — lobectomy for GGOs located in hilar regions
  Arms: lobectomy

SUMMARY:
GGO is a characteristic focus of early lung cancer. Due to the abundant peripheral blood vessels and bronchial tissues around the GGO lesions located in pulmonary hilar, only lobectomy could be used for the surgical treat of hilar GGO lesions which will make the significantly decline of the pulmonary function after surgery and affect the quality of life to a great extent. Our previous study has reported a new blunt-tip MWA electrode (MTC-3CA-II3, Vison Medical Inc.) for the treatment of GGO lesions. The blunt-tip MWA electrode could improve the safety of GGO ablation, significantly reduce the occurrence of bleeding and hemoptysis, which made it possible to ablate GGO in the hilar region safely. In this study, the blunt-tip MWA electrode was used in the treatment of patients with hilar GGO lesions, and the efficacy and safety of microwave ablation and lobectomy in the treatment of ground glass nodules located in the pulmonary hilar region were evaluated and compared.

ELIGIBILITY:
Inclusion Criteria:

1. The age ranged from 18 to 75 years old, male or female;
2. GGO lesions in the hilar region were diagnosed by imaging examination (CT / PET-CT). During the follow-up of 6-12 months, the lesions increased by more than 2mm, the solid components increased, or there were obvious solid components, or the GGOs were judged to be highly malignant by imaging.
3. The size of GGO lesions was 8mm-3cm, and the number of nodules was ≤ 3.
4. There was no lymph node metastasis, intrapulmonary metastasis or distant organ metastasis;
5. After multidisciplinary evaluation, the patients were feasible for lobectomy and CT guided microwave treatment;
6. No bleeding tendency, normal coagulation function or coagulation dysfunction can be corrected after treatment;
7. Patients and /or family members agreed to join the clinical trial and signed informed consent.

Exclusion Criteria:

1. The general condition of the patient is very poor, ECOG physical fitness score > 2, unable to tolerate lobectomy and MWA treatment, or has relevant contraindications;
2. The lesions had received other treatments before; patients with regional lymph node metastasis or distant metastasis or with pleural fluid and ascites;
3. Patients with poor compliance;
4. Severe heart, lung, kidney, brain and other important organ diseases;
5. The researcher believes that it is not suitable for inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year recurrence-free survival rate | 3 year after treatment
  3-year recurrence-free survival rate

SECONDARY OUTCOMES:
Postoperative hospital stay | During hospitalization
  Postoperative hospital stay
Total hospitalization expenses Total hospitalization expenses | During hospitalization
  Total hospitalization expenses
Incidence of complications | Within 1 month after operation
  Incidence of complications

IPD SHARING:
Plan to Share IPD: Undecided